CLINICAL TRIAL: NCT06550115
Title: Impact of Circulating and Tissue-specific Lipids on Vascular Function and Insulin Sensitivity in Chronic Night Shift Workers
Acronym: SHINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Josiane Broussard, Associate Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3717; R01HL168081 (NIH)
Record Dates: First submitted 2024-07-22; First posted 2024-08-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Circadian Rhythm Sleep Disorder of Shift Work Type; Metabolic Disease; Insulin Sensitivity; Blood Pressure
Keywords: Shift work; Sleep; Blood sugar; Metabolism; Lipids; Blood pressure
MeSH Terms: conditions — Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control eating during overnight work shift (Experimental): For 4 weeks, participants will eat during the biological night as is typically done in night shift workers.
  Interventions: Behavioral: Control eating
- Time-restricted eating during overnight work shift (Experimental): For 4 weeks, participants will refrain from eating during the biological night while maintaining the same sleep opportunity and daily energy intake and macronutrient distribution without changing 24h energy intake.
  Interventions: Behavioral: Time-restricted eating

INTERVENTIONS:
Behavioral: Time-restricted eating — Night shift workers will participate in 4 weeks of fasting during the biological nighttime while remaining awake during overnight work shifts.
  Other Names: Time-restricted feeding; TRF; TRE
  Arms: Time-restricted eating during overnight work shift
Behavioral: Control eating — Night shift workers will participate in 4 weeks of Control eating across the daytime and nighttime hours while remaining awake during overnight work shifts.
  Arms: Control eating during overnight work shift

SUMMARY:
People who experience repeated bouts of circadian misalignment, such as shift workers, are at higher risk of cardiovascular disease (CVD) and Type 2 diabetes (T2D) compared to daytime workers. However, the mechanism(s) by which shift work and associated circadian misalignment increase CVD and T2D risk are unknown. This project will examine whether elevated plasma lipids are a mechanism by which circadian misalignment impairs vascular function, insulin sensitivity, glucose homeostasis and muscle lipid accumulation, which could be targeted to prevent and treat cardiometabolic disease in people who chronically experience circadian misalignment, which includes more than 20% of the US workforce.

DETAILED DESCRIPTION:
There is growing recognition that timing of behaviors, such as eating, sleeping, and activity, have a significant impact on human health and disease risk. For example, when people are awake at the "wrong" time of the day (i.e. during the biological night), a mismatch occurs between behavior and biology, termed circadian misalignment. Shift workers experience repeated bouts of circadian misalignment and are at higher risk of cardiovascular disease (CVD) and Type 2 diabetes (T2D) compared to people who work days. However, the mechanism(s) by which shift work and associated circadian misalignment increase CVD and T2D risk are unknown.

Data from the investigators and others demonstrate impaired vascular endothelial function and insulin sensitivity during circadian misalignment, two important risk factors for future development of CVD and T2D. Furthermore, the investigators published and unpublished data support that circadian misalignment increases circulating bioactive lipids known to associate with impaired endothelial function and insulin resistance. Indeed, shift workers also have elevated circulating lipids, though it is not known which specific lipids are elevated, and whether they are associated with impaired vascular function and/or insulin sensitivity. Using a circadian-based eating intervention (time-restricted eating; TRE), we can consistently reduce lipids in circulation, as well as reduce heart rate and blood pressure and improve glucose homeostasis.

Therefore, the overall objective for this project is to examine whether increased plasma lipids are a potential mechanism by which chronic circadian misalignment impairs cardiovascular and metabolic health with the long-term goal of identifying novel therapeutic targets to combat the risks for disease when circadian misalignment is unavoidable. The central hypothesis is that reducing plasma lipids in night shift workers via TRE will improve vascular function, insulin sensitivity and glucose homeostasis, and reduce muscle tissue lipid accumulation. To test the hypothesis, we will conduct a 12-week randomized crossover study in 50 non-rotating night shift workers (25Females/25Males; 18-65years) with existing cardiometabolic risk factors. At the end of each 4-week outpatient condition (TRE vs Control with an intervening 4-week washout period), we will conduct rigorous 3-day inpatient assessment to determine the impact of plasma lipid reduction via TRE in chronic night shift workers on 1) vascular function and blood pressure; and 2) whole body and muscle-specific insulin sensitivity, glucose homeostasis and muscle lipid accumulation.

Achievement of these aims will identify a potential mechanism by which circadian misalignment impairs vascular function and insulin sensitivity (elevated plasma lipids), as well as a non-pharmacological tool (TRE) that could be implemented to reduce cardiometabolic disease risk in populations at elevated risk, in 20% of the US workforce who work nonstandard hours including military personnel, police, paramedics, firefighters, pilots, medical doctors and nurses, as well as people with sleep and circadian disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* worked the night shift for the last 1 year or more,
* habitually sleep 5-9 hours per 24h period (night shift workers typically experience chronic insufficient sleep),
* body mass index (BMI) of 20.0 - 35.0 kg/m2 and weight stable (plus or minus 5% of current body weight in the last 6 months); sedentary to mild physical activity level (less than 2 days of planned exercise per week);

Exclusion Criteria:

* existing diagnosed sleep or eating disorder (e.g. obstructive sleep apnea [OSA], periodic limb movements of sleep [PLMS], narcolepsy, travel more than 1 time zone in 3 weeks before the study; anorexia nervosa, more than one food allergy to maintain flexibility in diet planning);
* following any TRE (time-restricted eating) or intermittent fasting plan in the last year;
* following any special diet plan, like paleo, keto, gluten-free or vegan, that can affect the primary lipid outcome measures in the last 6 months; any clinically significant surgical condition within the last year;
* diagnosed diabetes or cardiovascular disease

  * The prevalence of insomnia in shift workers is fairly high, ranging from 12.8% to 76.4%, which is higher than estimated for the general population. Insomnia itself is associated with elevated neural cardiovascular responsiveness to stress compared to people without insomnia. Thus, since excessive sleepiness and symptoms of insomnia may be present in night shift workers they will not be exclusionary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure via 24-hour assessments | Collected during inpatient laboratory visit after 4 weeks of Control and TRE
  Four weeks of TRE during shift work will reduce 24-hour blood pressure versus Control.
Insulin sensitivity via clamp | Collected during inpatient laboratory visit after 4 weeks of Control and TRE
  Four weeks of TRE during shift work will improve insulin sensitivity versus Control.

SECONDARY OUTCOMES:
Cerebrovascular reactivity via transcranial doppler | Collected during inpatient laboratory visit after 4 weeks of Control and TRE
  Four weeks of TRE during shift work will improve cerebrovascular reactvity versus Control.
Muscle lipid accumulation via lipidomics | Collected during inpatient laboratory visit after 4 weeks of Control and TRE
  Four weeks of TRE during shift work will reduce muscle lipid accumulation versus Control.

OTHER OUTCOMES:
24-hour blood sampling for lipids, glucose, insulin, and vascular markers | Collected during inpatient laboratory visit after 4 weeks of Control and TRE
  Four weeks of TRE during shift work will improve 24-hour markers of vascular function versus Control.

CONTACTS AND LOCATIONS:
Overall Officials: Josiane L Broussard, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Josiane Broussard's Bibliography — http://www.ncbi.nlm.nih.gov/sites/myncbi/1JaM6qKzqsa5p/bibliography/45302103/public/?sort=date